CLINICAL TRIAL: NCT00192946
Title: Cardiac Resynchronization Therapy (CRT) in the Early Phase After Heart Surgery
Brief Title: The CRT-KIR Study (Cardiac Resynchronization Therapy [CRT] in the Early Phase After Heart Surgery)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study population is smaller than expected. No subjects were included.
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF 01-230/04
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2006-02

CONDITIONS: Bundle-Branch Block
Keywords: Cardiac resynchronization; Heart failure; open heart surgery; surgery
MeSH Terms: conditions — Bundle-Branch Block; Heart Failure

INTERVENTIONS:
Procedure: Temporary cardiac resynchronization therapy

SUMMARY:
In patients with broad QRS complexes on electrocardiogram (ECG), the delayed electrical activation of the left heart chamber will cause abnormal contraction.This has been shown to be possible to treat by a special pacemaker treatment which includes pacing of the left heart chamber (= CRT treatment).

In this study the researchers will investigate the effect of acute CRT treatment in the early phase after open heart surgery.

DETAILED DESCRIPTION:
Patients with bundle branch block have a delayed electrical activation of the left ventricle causing abnormal contractility of the left ventricle.

We hypothesize that patients may benefit from short term (= 72 hours) CRT (Cardiac Resynchronization Therapy) in the early phase after open heart surgery.

Patients: reduced LV function and bundle branch block.

Study type: randomisation to CRT versus standard postoperative treatment

Study variables: cardiac output, echocardiographic measures, p-BNP and hours with inotropic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for open heart surgery (coronary artery bypass graft [CABG] or mitral valve surgery or aortic valve surgery or combinations of the above mentioned surgical procedures) and LV ejection fraction < 35% and bundle branch block (QRS > 9.12 s)

Exclusion Criteria:

* Severe right heart failure
* Permanent atrial fibrillation
* Congenital heart disease
* Serious non-cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Study Completion 2008-09 (Estimated)

PRIMARY OUTCOMES:
Non invasive cardiac output after 72 hours CRT (versus control) treatment

SECONDARY OUTCOMES:
Echocardiographic measures of left ventricular (LV) function
Mixed venous oxygen saturation
Invasively determined cardiac output
Plasma brain natriuretic peptide (p-BNP)
Number of hours with inotropic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Svendsen, MD, Principal Investigator — Rigshospitalet, Denmark